CLINICAL TRIAL: NCT06709170
Title: Safety & Efficacy of a Novel Asymmetrical Linear Stapler (NALS) for Securing Distal Resection Margin in Laparoscopic Rectal Cancer Surgery: Pilot Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Seoul National University Boramae Hospital (Other); National Cancer Center, Korea (Other Government); Kyungpook National University Chilgok Hospital (Other)
Responsible Party: Principal Investigator, Ryoo, Seung-Bum, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-3198
Record Dates: First submitted 2024-11-17; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Colo-rectal Cancer
Keywords: Rectal cancer; Frozen sections; Margins of Excision
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Margins of Excision

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Novel asymmetrical linear stapler (Experimental): Rectal cancer patients randomized to this group will use the novel asymmetrical linear stapler for distal rectum transection, and with 2 rows of stapler lines instead of 3, sufficient tissue is left on the specimen side to harvest the true distal margin for accurate pathological evaluation.
  Interventions: Device: Novel asymmetrical linear stapler
- Control (Active Comparator): Rectal cancer patients in the control group will use the conventional Signia™ stapler (Medtronic co.) as routinely used in the centers involved with the study, which has triple stapling technology (3 rows of stapler lines on both sides of transection)
  Interventions: Device: Signia™

INTERVENTIONS:
Device: Novel asymmetrical linear stapler — Novel asymmetrical linear stapler
  Arms: Novel asymmetrical linear stapler
Device: Signia™ — Signia™
  Arms: Control

SUMMARY:
Through the use of a novel asymmetrical linear stapler (NALS, Meditulip co. Ltd.), we aim to prove that true distal margins greater than 1cm may be harvested more readily and easily compared to the conventional staplers. The study is designed as a pilot RCT of 30 patients in each group, with the primary outcome of distal margin length >1cm. Secondary outcomes include anastomosis dehiscence and time taken to harvest the distal margin.

DETAILED DESCRIPTION:
Current evidence indicates distal margins of greater than 1cm from the tumor is necessary for superior oncologic outcomes. In middle to lower rectal cancer, where the tumor is close to the anus, sparing the anus whilst securing such a margin may prove difficult.

Failure to secure sufficient margin length may end up in cancer recurrence, but inaccurate assessment of the margin status may also cause further unnecessary resection or failure to spare the anus.

The novel asymmetrical linear stapler was designed specifically with this problem in mind, and one row of stapling was removed from the specimen side to allow easier harvesting of a undisrupted distal margin tissue for pathological evaluation.

This study is a pilot RCT of 30 patients each in the novel stapler group and control group, to prove the non-inferiority in safety and superiority in harvesting the distal margin (assessed by length of margin and time to harvest).

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer patients between the age of 19~79, who require anus preserving laparoscopic rectum resection surgery

Exclusion Criteria:

* Advanced rectal cancer that invades surrounding structures or has known distant metastasis
* Uncontrolled comorbidities
* Patients otherwise considered unsuitable for the study

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
True distal margin length > 1cm | Intraoperative
  True distal margin: The length of tissue from the distal edge of the specimen to the distal tumor margin in the surgical specimen

SECONDARY OUTCOMES:
Early anastomosis leakage | From randomization until the date of first documented sign of leakage, assessed up to 30 days
  Anastomosis leakage within 30 days of surgery will be documented and reported as an outcome. The International Study Group of Rectal Cancer definition of anastomosis leakage will be used to define the outcome (defect of the intestinal wall at the anastomotic site leading to a communication between the intra- and extraluminal compartments, requiring NPO or other intervention).
  Patients that have clinical signs of infection (fever, sepsis, inflammatory lab change or abdominal drain color change) with either fluid collection near the anastomosis or an anastomosis defect on CT imaging will be diagnosed as having anastomosis leakage. CT scans will not be taken routinely, but will be performed when signs of infection (such as abdominal tenderness or high fever) are present.
  Severity of the anastomosis leak will be graded according to the International Study Group of Rectal Cancer grading system (grade A, B, C) depending on the necessary intervention (none, non-surgical or surgical).
Time to harvest margin | Intraoperative (from the beginning of frozen section specimen harvest until the acquirement is completed. This process will be timed by a member of the surgical team using a timer.)
  Time (seconds) taken to harvest the distal margin from the specimen for frozen section biopsy
Specimen integrity | Intraoperative (at the time point of the frozen section pathology report)
  The pathologist evaluation of whether the whole thickness of bowel was harvested in the distal margin frozen section biopsy. This will be requested and reviewed, reported in the final pathologist report.
Sphincter preservation rate | From randomization until the end of clinical data collection, assessed up to 120 days.
  Although all eligible candidates will be planned for sphincter-preserving surgery, there are some cases where the distal margin is not suffice for an R0 resection and thus receive non-sphincter preserving surgery. The incidence of such non-sphincter preserving surgery (example: abdominoperineal resection) will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongro-gu, South Korea

IPD SHARING:
Plan to Share IPD: No